CLINICAL TRIAL: NCT02961192
Title: Using Social Incentives and Patient-Generated Health Data to Change Health Behaviors and Improve Glycemic Control Among Type 2 Diabetics
Brief Title: Social Incentives to Improve Diabetes
Acronym: iDiabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 825372
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Type II; Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will receive a wireless weight scale and a wearable activity tracker to monitor their weight and step counts.
- Supportive (Experimental): Participants will receive a wireless weight scale and a wearable activity tracker to monitor their weight and step counts. Additionally, participants will play a game designed with insights from behavioral economics. The game will involve points and levels. In addition to playing the game, participants will identify a family member or friend to receive updates and support them in their progress.
  Interventions: Behavioral: Supportive social incentive
- Competitive (Experimental): Participants will receive a wireless weight scale and a wearable activity tracker to monitor their weight and step counts. Additionally, participants will play a game designed with insights from behavioral economics. The game will involve points and levels. In this arm, participants will be placed into competitive groups with one or two other participants to play the game.
  Interventions: Behavioral: Competitive social incentive
- Collaborative (Experimental): Participants will receive a wireless weight scale and a wearable activity tracker to monitor their weight and step counts. Additionally, participants will play a game designed with insights from behavioral economics. The game will involve points and levels. In this arm, participants will be placed into collaborative groups with one or two other participants to play the game.
  Interventions: Behavioral: Collaborative social incentive

INTERVENTIONS:
Behavioral: Supportive social incentive — A family member or friend will be used as a support person in this study, to receive updates and support the participant in their progress.
  Arms: Supportive
Behavioral: Competitive social incentive — Participants in this intervention will be competing against each other in the game.
  Arms: Competitive
Behavioral: Collaborative social incentive — Participants in this intervention will be working with each other in the game.
  Arms: Collaborative

SUMMARY:
In this study, we will conduct a one-year, four-arm, randomized, controlled trial to compare three social incentive-based gamification interventions to control for promoting physical activity and weight loss toward improved glycemic control among type 2 diabetics.

DETAILED DESCRIPTION:
This is a four-arm, one-year randomized, controlled trial. The study will be conducted using Way to Health, an automated information technology platform at the University of Pennsylvania that integrates wireless devices, conducts clinical trial randomization and enrollment processes, delivers messaging (text or email) delivers self-administered surveys, automates payment transfers, and securely captures data for research purposes.

The study team will identify potential participants from the electronic health record at the University of Pennsylvania Health System. Interested participants will be instructed to visit the study website to create an account, review and complete informed consent, and complete an eligibility survey. Eligible participants will be instructed to obtain a hemoglobin A1c and LDL-C laboratory test. If the hemoglobin A1c is 8.0 or greater and the participant is still interested in continuing the enrollment process, a wearable activity tracking device will be mailed to them. After that, the participant will be scheduled for an in-person visit with the study team to complete the enrollment process.

Participants will be randomly assigned in blocks of four groups to one of the four study arms stratified based on whether the group of individuals already knew each other or not. Groups will have three individuals unless the individuals were already socially connected prior to the study, in which case they will be allowed to be randomized as a group of two or three. Participants randomized to the control arm will receive no other interventions.

Each participant in the intervention arms will be asked to choose their goals for the study as follows: 1) Choose a weight loss goal that is 6%, 7%, or 8% of their baseline weight rounded up to the next pound; 2) Choose a daily step count goal that is 33%, 40%, or 50% greater than their baseline rounded up to the nearest hundred, or choose their own step goal as long as it is at least 1500 steps above their baseline; 3) Choose a HbA1c reduction goal of 1.5%, 2%, or 2.5%.

Participants in arms 2-4 will be entered into an intervention approach that has points and levels designed to incorporate insights from behavioral economics. On a daily basis, they will be asked to weigh-in. They will have a weekly weight target and mean step goal. Weekly feedback will differ among the three arms to induce the different social incentives.

The primary outcome variables are change in mean daily steps, weight in pounds, and hemoglobin A1c from baseline to end of the one-year study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 70 years
2. Ability to read and provide informed consent to participate in the study
3. Diagnosis of type 2 diabetes with a hemoglobin A1c of 8.0 or greater
4. Self-reported body mass index (BMI) of 25 or greater.
5. Smartphone or tablet compatible with the application for the wearable activity tracking device and wireless weight scale.

Exclusion Criteria:

1. Conditions that would make participation infeasible such as inability to provide informed consent, illiteracy or inability to speak, read, and write English
2. Conditions that would make participation unsafe such as pregnancy, previous diagnosis of an eating disorder, or history of unsafe weight loss practices
3. Already enrolled in another study targeting physical activity, weight loss, or glycemic control
4. Any other medical conditions or reasons he or she is unable to participate in the study for one year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | 12 months
  Change in hemoglobin A1c from baseline to the end of the one-year study.
Change in weight in pounds | 12 months
  Change in weight in pounds from baseline to the end of the one-year study.
Change in mean daily steps | 12 months
  Change in baseline step count compared to the entire one-year study period.

SECONDARY OUTCOMES:
Change in mean daily steps | 6 months
  Change in baseline step count compared to the first 6 months of the study period
Change in weight in pounds from baseline to the study midpoint | 6 months
  Change in weight from baseline to the six-month midpoint of the study
Change in hemoglobin A1c from baseline to the study midpoint | 6 months
  Change in hemoglobin A1c to the six-month midpoint of the study
Change in LDL-C levels | 6 months
  Change in LDL-C from baseline to the six-month midpoint of the study
Change in LDL-C levels | 12 months
  Change in LDL-C from baseline to the end of the one-year study.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Patel MS, Small DS, Harrison JD, Hilbert V, Fortunato MP, Oon AL, Rareshide CAL, Volpp KG. Effect of Behaviorally Designed Gamification With Social Incentives on Lifestyle Modification Among Adults With Uncontrolled Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e2110255. doi: 10.1001/jamanetworkopen.2021.10255. PMID 34028550
- [Derived] Fortunato M, Harrison J, Oon AL, Small D, Hilbert V, Rareshide C, Patel M. Remotely Monitored Gamification and Social Incentives to Improve Glycemic Control Among Adults With Uncontrolled Type 2 Diabetes (iDiabetes): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 20;8(11):e14180. doi: 10.2196/14180. PMID 31746765